CLINICAL TRIAL: NCT06191848
Title: Effect of Subcutaneous Tirzepatide Once-weekly in Patients With Obesity and Knee Osteoarthritis (STOP KNEE-OA): A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Subcutaneous Tirzepatide Once-weekly in Patients With Obesity and Knee Osteoarthritis (STOP KNEE-OA)
Acronym: STOP KNEE-OA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 75430
Record Dates: First submitted 2023-12-18; First posted 2024-01-05 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Knee Osteoarthritis; Osteoarthritis, Knee
Keywords: Osteoarthritis; Obesity; Total knee replacement
MeSH Terms: conditions — Obesity; Osteoarthritis, Knee; Osteoarthritis | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tirzepatide (Experimental): Drug: Tirzepatide is a glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide-1receptor (GLP1R) agonist Dose: Tirzepatide will be initiated at 2.5mg once weekly, with the dose increasing by a further 2.5mg every four weeks until the target weekly dose of 15mg is achieved (or participants reach a lower maximum tolerated dose of 5mg or 10mg).
  Duration: 72-weeks Mode: subcutaneous
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Drug: Placebo Dose: once-weekly Duration: 72 weeks Mode: subcutaneous
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Participants will receive tirzepatide subcutaneously
  Arms: Tirzepatide
Drug: Placebo — Participants will receive placebo subcutaneously
  Arms: Placebo

SUMMARY:
This is a trial of tirzepatide in people with obesity and knee osteoarthritis. The main purpose of this study is to see if tirzepatide can reduce number of these participants who require a knee replacement. Participants will be randomized to take a weekly injection of tirzepatide or a placebo for a total of 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index of ≥ to 30 kg/m2.
* Report one or more previous unsuccessful attempt to lose body weight via lifestyle modification.
* Have been deemed eligible to enter the waiting list for primary knee replacement for the treatment of osteoarthritis in the target joint by an orthopaedic surgeon at one of the participating study sites.
* Have moderate-to-severe knee osteoarthritis in the target joint, defined as a Kellgren-Lawrence grade two or greater.
* Be willing to and capable of learning how to self-inject the study drug and follow study procedures for the duration of the trial.
* Provide informed consent to study participation in line with the requirements of the human research ethics committee of the study site.

Female participants must:

* Not be currently pregnant or breastfeeding AND
* Not be of reproductive potential, defined as:
* Infertile due to surgical sterilization or congenital anomaly, OR
* Post-menopausal defined as:
* A woman over the age of 40 years with spontaneous cessation of menses for at least 12 consecutive months (in the absence of medications known to induce amenorrhea), with a follicle-stimulating hormone ≥40mIU/mL, and a negative pregnancy test prior to study entry, OR
* A woman over the age of 55 years with cessation of menses for at least 12 consecutive months (in the absence of medications known to induce amenorrhea), OR
* A woman over the age of 55 years that has commenced hormone replacement therapy after a documented diagnosis of menopause.

Exclusion Criteria:

Participant will be ineligible for inclusion if they meet any of the following criteria:

* Have been deemed eligible to enter the waiting list for knee replacement in the contralateral knee by an orthopaedic surgeon at one of the participating study sites.
* Have used any prescription medications intended to promote weight loss (e.g., tirzepatide, liraglutide, semaglutide) in the three months prior to screening.
* Have previously undergone any surgical or endoscopic procedure intended to promote weight loss.
* Have been diagnosed with type 1 diabetes mellitus (T1DM) or T2DM
* Have laboratory evidence indicative of diabetes mellitus during screening.
* Have personal or family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
* Have an active malignancy (excluding basal or squamous cell skin cancer).
* Have had a transplanted organ or awaiting an organ transplant
* Have received chronic systemic glucocorticoid therapy (for more than 14 days) in prior 3 months or have a significant, active autoimmune abnormality (e.g., lupus or rheumatoid arthritis) that the study doctor deems likely to require systemic glucocorticoid therapy during the next 18 months.
* Have any other medical conditions, abnormal laboratory tests or concomitant medications that make them unsuitable for participation:

  * Have a clinically significant gastric emptying abnormality.
  * Have had a history of acute or chronic pancreatitis.
  * Have obesity induced by other endocrinologic disorders
  * Have an unstable psychiatric disorder
  * Have a Patient Health Questionnaire (PHQ-9) score of >15 during screening
  * Have been deemed by the study doctor to be actively suicidal,
* Have answered "yes" to questions 4 or 5 on the "Suicidal Ideation" section of the Columbia-Suicide Severity Rating Scale (C-SSRS) during screening, OR
* Have answered yes to any questions in the "Suicidal Behaviour" section of the C-SSRS during screening. AND
* The behaviour or ideation occurred in the last month

  * Have uncontrolled hypertension (systolic blood pressure above or equal to 160 mmHg and/or diastolic blood pressure above or equal to 100 mmHg)
  * Have had within the past 6 months prior to randomisation any of the following: acute myocardial infarction, cerebrovascular accident, unstable angina, or hospitalisation due to congestive cardiac failure (are also exclusion criteria for elective knee replacement)
  * Have severe renal impairment defined as an eGFR <30 mL/min/1.73 m2 at screening visit.
  * Have thyroid-stimulating hormone outside of the range of 0.4 to 6.0 mIU/L at screening visit
  * Have acute or chronic hepatitis or abnormal liver function tests as measured by either alanine aminotransferase or alkaline phosphatase >200 IU.
  * Have any other known contraindication to any glucagon-like peptide-1 receptor agonists.
* Are study site personnel, or immediate family of a member of the study site.
* Have been enrolled in any other study of an investigational product within the past ninety days or are currently enrolled in such a study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2037-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who undergo knee replacement in the target joint | within 72 weeks of randomization
  Percentage of patients who undergo knee replacement in the target joint

SECONDARY OUTCOMES:
Osteoarthritis Pain | Baseline, Week 72
  Change from Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score. The WOMAC Pain subscale has 5-items, with a possible score range of 0-20, with higher scores indicating worse pain.
Osteoarthritis Function | Baseline, Week 72
  Change from Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Function Subscale Score. The WOMAC Function subscale has 17-items, with a possible range of 0-68, with higher scores indicating worse functional impairment.
Osteoarthritis Stiffness | Baseline, Week 72
  Change from Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score. The WOMAC Stiffness subscale has 2-items, with a possible range of 0-8, with higher score indicating worse stiffness.
Percentage change in bodyweight | Baseline, Week 72
  Mean percentage change in body weight at 72 weeks after randomization
≥5% body weight reduction | Baseline, Week 72
  Percentage of participants with ≥5% body weight reduction at 72 weeks after randomization
≥10% body weight reduction | Baseline, Week 72
  Percentage of participants with ≥10% body weight reduction at 72 weeks after randomization
≥20% body weight reduction | Baseline, Week 72
  Percentage of participants with ≥20% body weight reduction at 72 weeks after randomization
Physical Health | Baseline, Week 72
  Mean change in the 36-item Short Form (SF-36) Physical Component Summary at 72 weeks after randomization. The SF-36 Physical Component Summary, a lower score indicates poorer physical health.
Mental Health | Baseline, Week 72
  Mean change in the 36-item Short Form Survey (SF-36) Mental Component Summary at 72 weeks after randomization. For the SF-36 Mental Component Summary, a lower score indicates poorer mental health.
Physical Activity | Baseline, Week 72
  Mean change in Physical Activity Scale for the Elderly (PASE) score at 72 weeks after randomization. The PASE has 12-items with a total score range from 0-400 or more, with higher scores indicating greater physical activity.
Non-opioid prescription pain medication use | Baseline, between 68-72 weeks
  Proportion of participants reporting use of non-opioid prescription analgesics between 68-72 weeks after randomization
Opioid prescription pain medication use | Baseline, between 68-72 weeks
  Proportion of participants reporting use of prescription opioid analgesics between 68-72 weeks after randomization
Mean change in use of prescription opioid pain medication | Baseline, between 68-72 weeks
  Mean change in prescription opioids dose at 72 weeks after randomization
Participant willingness to undergo knee replacement surgery | within the 72 weeks since randomization
  Proportion of patients who undergo knee replacement in the target joint within 72 weeks of randomization or re-enter the waiting list within 72 weeks of randomization.
Long-term (5-year) progression to knee replacement | within 260 weeks of randomization
  Percentage of patients who undergo knee replacement in the target joint within 5-years
Long-term (10-year) progression to knee replacement | within 520 weeks of randomization
  Percentage of patients who undergo knee replacement in the target joint within 10-years

CONTACTS AND LOCATIONS:
Overall Officials: Michelle M Dowsey, Principal Investigator — University of Melbourne
Locations (4):
- Australia (4):
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Western Health, Melbourne, Victoria
  - Austin Health-Repatriation Hospital, Melbourne, Victoria
  - Eastern Health, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval by the principal investigator of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary results publication. Data will be indefinitely available for requesting
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-02-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT06191848/SAP_000.pdf